CLINICAL TRIAL: NCT07229456
Title: Evaluation of the Role of N Acetyl Cysteine and Vitamin D in Improving Outcomes After Corrosive Ingestion
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: FAMSU MS 611/2024
Record Dates: First submitted 2025-09-05; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Corrosive Injury
Keywords: corrosive ingestion; vitamin D; N acetyl cysteine
MeSH Terms: interventions — Acetylcysteine; Cholecalciferol; Control Groups

STUDY DESIGN:
Intervention Model Description: Eighty patients were randomly assigned into four groups (1 control and 3 intervention groups 20 patients each)
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control (Active Comparator): Patients allocated in this group will receive the standard treatment protocol only according to PCC-ASUH guidelines
  Interventions: Drug: control group
- N acetyl cysteine group (Active Comparator): * Patients in this group received the standard treatment protocol according to PCC-ASUH guidelines in addition to NAC with loading dose of 150 mg/kg diluted in 200 ml dextrose 5% or saline over 1 hour, followed by a maintenance dose of 50 mg/kg diluted in 500 ml of dextrose 5% or saline over 4 hours then followed by 100 ml/kg diluted in 1000 ml of dextrose 5% or saline over 16 hours
  * Preparation and administration of NAC were adjusted according to the age of the patient. In those >12 years old, total volume (NAC and IV fluid) for the bolus, 4-hour infusion, and 16 hours infusion was 200 ml, 500 ml, and 1 liter, respectively. In children <12 years but over 20 kg, volumes were 100 ml, 250 ml, and 500 ml respectively. In those under 20 kg volumes were 3 ml/kg, 7 ml/kg, and 14 ml/kg respectively
  Interventions: Drug: N Acetyl Cysteine; Drug: control group
- vitamin D group (Active Comparator): Patients in this group received the standard treatment protocol according to PCC-ASUH guidelines in addition to vitamin D in a single intramuscular high-dose (300,000 IU) which was given to all patients regardless patient's age
  Interventions: Drug: Vitamin D (Cholecalciferol ); Drug: control group
- N acetyl cysteine and Vitamin D group (Active Comparator): Patients in this group received the standard treatment protocol according to PCC-ASUH guidelines in addition to both vitamin D and NAC, in the same doses as groups (2 and 3).
  Interventions: Drug: N Acetyl Cysteine; Drug: Vitamin D (Cholecalciferol ); Drug: control group

INTERVENTIONS:
Drug: N Acetyl Cysteine — N-acetyl cysteine (NAC) has a well-established safety profile, its remarkable antioxidant and anti-inflammatory capacity is the biochemical basis used to treat several diseases related to oxidative stress and inflammation. The primary role of NAC as an antioxidant stems from its ability to increase the intracellular concentration of glutathione (GSH), which is responsible for cellular redox imbalance .
  It is assumed that NAC acts as a reductant of disulfide bonds, a scavenger of reactive oxygen species and/or a precursor for glutathione biosynthesis N-acetyl cysteine was observed to be useful in the treatment of esophageal damage associated with corrosive substances and in achieving histopathological improvement in an experimental setting
  Other Names: Acetyle cysteine; Hidonac
  Arms: N acetyl cysteine and Vitamin D group; N acetyl cysteine group
Drug: Vitamin D (Cholecalciferol ) — counteracts the pro-fibrotic signals, such as transforming growth factor-β1 (TGF-β1), through several biochemical mechanisms. This inhibits myofibroblasts activation and extra cellular matrix deposition. In addition, vitamin D reduces the expression of pro-fibrotic target genes The antioxidant effect of vitamin D is between the newest suggested non-calcemic roles of this compound through inducing the expression of several molecules involved in the antioxidant defense system including glutathione, glutathione peroxidase and superoxide dismutase (SOD) and suppressing the expression of NADPH oxidase
  Other Names: (Cholecalciferol ); osavidin
  Arms: N acetyl cysteine and Vitamin D group; vitamin D group
Drug: control group — Patients allocated in this group received the standard treatment protocol only according to PCC-ASUH guidelines.

SUMMARY:
The goal of this clinical trial is to learn if N acetyl cysteine and vitaminD work to improve outcomes after corrosive ingestion in children.

The main questions it aims to answer are:

Does N acetyl cysteine and vitamin D decrease incidence of strictures after corrosive ingestion in children.

Researchers will compare the effect of N acetyl cysteine and vitamin D in decreasing complication , length of hospital stay and start of complete oral intake Eighty patients were randomly assigned into four groups (1 control and 3 intervention groups 20 patients each)

Group 1 (Control group):

o Patients allocated in this group received the standard treatment protocol only according to PCC-ASUH guidelines

Group 2 (NAC group):

o Patients in this group received the standard treatment protocol according to PCC-ASUH guidelines in addition to NAC with loading dose of 150 mg/kg diluted in 200 ml dextrose 5% or saline over 1 hour, followed by a maintenance dose of 50 mg/kg diluted in 500 ml of dextrose 5% or saline over 4 hours then followed by 100 ml/kg diluted in 1000 ml of dextrose 5% or saline over 16 hours

Group 3 (Vitamin D group):

Patients in this group received the standard treatment protocol according to PCC-ASUH guidelines in addition to vitamin D in a single intramuscular high-dose (300,000 IU) which was given to all patients regardless patient's age

Group 4 (NAC+Vitamin D group):

Patients in this group received the standard treatment protocol according to PCC-ASUH guidelines in addition to both vitamin D and NAC, in the same doses as groups (2 and 3

DETAILED DESCRIPTION:
The current study is a controlled randomized, single-blinded clinical trial, conducted on acutely poisoned patients with confirmed history of corrosive ingestion who were admitted to the Poison Control Center, Ain Shams University Hospitals (PCC-ASUH) The required sample size is 80 patients, 20 patients in each group according to the recommendation of statistics committee (Community Medicine, Environmental, and Occupational Medicine Department - Faculty of Medicine, Ain shams University)

Eighty patients were randomly assigned into four groups (1 control and 3 intervention groups 20 patients each)

Group 1 (Control group):

o Patients allocated in this group received the standard treatment protocol only according to PCC-ASUH guideline This included patient stabilization, maintaining patent airways, oxygen administration and ventilatory support when necessary.

In patients presenting with oral symptoms such as lip edema, excessive drooling (sialorrhea), or oral ulcers, the child was kept NPO to prevent further irritation. Topical treatments including antibiotics, anti-inflammatory agents, and antifungals were applied to manage local infection and inflammation.

Intravenous fluids were started to maintain hydration, with the volume calculated based on the Holliday-Segar method as follows: 100 mL/kg for the first 10 kg of body weight, 50 mL/kg for the next 10 kg, and 20 mL/kg for any weight above 20 kg. Fluid selection depended on the clinical condition where isotonic fluids such as 0.9% saline were often used initially, followed by hypotonic solutions containing dextrose and electrolytes for maintenance to prevent complications like hyponatremia or fluid overload Corticosteroids, especially dexamethasone, were administered when there was severe lip edema or suspected airway swelling to reduce inflammation and to prevent airway compromise. The typical dose used was 0.6 mg/kg, up to a maximum of 10 mg. However, steroids were avoided in children presenting with hematemesis or melena, due to the risk of worsening gastrointestinal bleeding.

In cases with GIT symptoms, supportive care was provided. If vomiting was present, ondansetron was administered at a dose of 4 mg every 8 hours until symptoms were controlled, and then on demand. To treat esophagitis and abdominal discomfort, proton pump inhibitors (PPIs) such as omeprazole were used to reduce acid secretion and promote healing of the mucosa. Omeprazole was given at 0.4-0.8 mg/kg, either every 12 or 24 hours, depending on symptom severity.

For children with signs of upper GI bleeding such as hematemesis or melena, urgent resuscitation was initiated. This included blood transfusion in cases of hemoglobin drop, fresh frozen plasma, IV PPI infusion, and hemostatic agents like tranexamic acid (Kapron), etamsylate (Dicynone), and vitamin K (Konakion). Diagnostic imaging such as chest X-ray, erect and supine abdominal X-rays, and abdominal ultrasound were performed to assess complications like perforation or effusion.

In children with respiratory symptoms, especially those with stridor or laryngeal edema, adrenaline was administered to reduce airway swelling. If chemical pneumonitis was suspected, inhaled bronchodilators (e.g., salbutamol every 4-6 hours), mucolytics like N-acetyl cysteine (NAC) or hypertonic saline every 6 hours, and antibiotics (based on culture and sensitivity) were given. Additionally, IV paracetamol at 10-15 mg/kg every 6 hours was used for fever, pain, and inflammation.

For patients who developed dysphagia and could not tolerate oral or enteral feeding for more than 3-5 days, total parenteral nutrition (TPN) was initiated to prevent malnutrition and support tissue healing. TPN was carefully tailored to the child's age, weight, and clinical status. Fluid needs were typically 100-150 mL/kg/day. Glucose, the main energy source, was started at 6-8 mg/kg/min in neonates (up to 12-14 mg/kg/min as tolerated) and 5-10 mg/kg/min in older children. Amino acids, essential for growth and repair, were given at 2-3 g/kg/day in neonates and 1-2 g/kg/day in older children. Lipids were started early at 1-2 g/kg/day, increasing to 3 g/kg/day if needed, particularly in neonates.

Electrolyte supplementation was guided by lab values: sodium (2-5 mEq/kg/day), potassium (1-3 mEq/kg/day), calcium (50-100 mg/kg/day of elemental calcium), magnesium (0.25-0.5 mEq/kg/day), and phosphate (1-2 mmol/kg/day). Micronutrients were also essential - daily multivitamins were given (e.g.,1 mL/day for infants, 2-5 mL/day for older children), along with trace elements such as zinc (100-400 mcg/kg/day), copper (20 mcg/kg/day), manganese (1 mcg/kg/day), selenium (2 mcg/kg/day), and chromium (0.14-0.2 mcg/kg /day).

Group 2 (NAC group):

o Patients in this group received the standard treatment protocol according to PCC-ASUH guidelines in addition to NAC with loading dose of 150 mg/kg diluted in 200 ml dextrose 5% or saline over 1 hour, followed by a maintenance dose of 50 mg/kg diluted in 500 ml of dextrose 5% or saline over 4 hours then followed by 100 ml/kg diluted in 1000 ml of dextrose 5% or saline over 16 hours

Preparation and administration of NAC were adjusted according to the age of the patient. In those>12 years old, total volume (NAC and IV fluid) for the bolus, 4-hour infusion, and 16 hours infusion was 200 ml, 500 ml, and 1 liter, respectively. In children <12 years but over 20 kg, volumes were 100 ml, 250 ml, and 500 ml, respectively. In those under 20 kg, volumes were 3 ml/kg, 7 ml/kg, and 14 ml/kg, respectively

Group 3 (Vitamin D group):

Patients in this group received the standard treatment protocol according to PCC-ASUH guidelines in addition to vitamin D in a single intramuscular high-dose (300,000 IU) which was given to all patients regardless patient's age

Group 4 (NAC + Vitamin D group):

Patients in this group received the standard treatment protocol according to PCC-ASUH guidelines in addition to both vitamin D and NAC, in the same doses as groups (2 and 3)

Study tools:

Data collection:

A sheet will be constructed for every patient including the following collected data:

(a) History taking:

* Socio-demographic data:
* These include data regarding age, sex, and residence. (b) Intoxication data:
* Type of corrosive substance (acid or alkali).
* Manner of poisoning, whether suicidal, accidental, or criminal.
* Time elapsed between corrosive ingestion and arrival to PCC-ASUH (Delay time).
* Past medical history. (b) Clinical examination
* General examination:

  o Vital data including blood pressure, pulse, respiratory rate, and temperature.
* Systemic examination:

  * Chest and abdominal examination
  * Symptoms (e.g., lip edema, tongue ulcers, vomiting, dysphagia, salivation, and others).

(C) Investigations:

I) Laboratory investigations:

Both arterial and venous blood samples will be obtained, under complete aseptic condition, for performing the following investigations on admission, 24 hours, and 48 hours after receiving the treatment.

* Arterial blood gas analysis.
* Random blood glucose.
* Serum electrolytes (sodium and potassium).
* Liver enzymes (ALT and AST).
* Renal function tests (Serum urea and creatinine).
* Complete blood count. The neutrophil to lymphocyte ratio and the platelet to lymphocyte ratio will be calculated by dividing the absolute count of neutrophils and platelets, respectively, over the absolute count of lymphocytes (Siddique et al., 2021).
* C-reactive protein (CRP).

II) Radiological investigations:

* Plain chest and abdominal radiograph will be carried out at the time of admission.
* Barium swallow and meal will be done 21 days after acute corrosive ingestion.

ELIGIBILITY:
Inclusion Criteria:

* The study included all patients aged from 0 to 18 years old, of both sex, admitted to the PCC-ASUH with confirmed history of corrosive ingestion and exhibiting moderate or severe symptoms (as determined by Poisoning Severity Score 2 or 3, respectively) and DROOL score (Drooling, Reluctance, Oropharynx, Others, and leukocytosis) ≤ 6

Exclusion Criteria:

* o Asymptomatic patients.

  * Patients exposed to corrosives through routes other than ingestion (e.g., inhalation, dermal or eye contact).
  * Patients with a delay time of more than 24 h.
  * Patients who co-ingested other poisons.
  * Patients presented with GIT perforation after corrosive ingestion.
  * Patients who received treatment before admission.
  * Patients receiving chemotherapy or radiation.
  * Patients with known blood disorders or malignancy.
  * Patients with history of blood transfusion in the last 90 days.
  * Patients with recent infections in the last 14 day

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Stricture formation | 21 days after corrosive ingestion
  Stenosis of esophygeal lumen or gastric lumen after corrosive ingestion which will be seen in barium swallow and meal

CONTACTS AND LOCATIONS:
Overall Officials: Eglal H Elawady, Professor of toxicology, Study Chair — faculty of medicine - Ain Shams University; Walaa G Abdelhamid, Assistant Professor, Study Chair — faculty of medicine - Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol